CLINICAL TRIAL: NCT00143624
Title: Effect of Rosiglitazone Maleate (Avandia®) on Carotid Intima Media Thickness, Brachial Artery Reactivity, Glucose Metabolism, Blood Lipid Concentrations, Body Fat Distribution, and Biochemical Markers of Cardiovascular Risk in Patients With the HIV Metabolic Syndrome
Brief Title: Rosiglitazone (Avandia®) Treatment in HIV: Its Effect on Blood Vessels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Dr. Greg Bondy, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02-0086; CTN 178
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Atherosclerosis; HIV Infections
Keywords: Treatment Experienced; HIV Metabolic Syndrome; Atherosclerosis in HIV
MeSH Terms: conditions — Atherosclerosis; HIV Infections | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): The first group will receive 8 mg of the study drug (rosiglitazone).
  Interventions: Drug: Rosiglitazone maleate
- 2 (Placebo Comparator): The second group will be given a placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosiglitazone maleate — See Detailed Description.
  Arms: 1
Drug: Placebo — See detailed description.
  Arms: 2

SUMMARY:
This trial will study the effect of rosiglitazone on the progression of atherosclerosis (hardening of blood vessels) through improvements of the sugar and fat metabolism (body buildup, breakdown and excretion of sugar and fat).

Participants will be randomly assigned to one of two groups: the first group will receive 8 mg of the study drug and the second group will be given a placebo, though neither group will know which formulation they are receiving. The study will follow both groups for one year, during which it will measure changes in blood vessel composition and activity, sugar metabolism, concentration of blood fat, and body fat distribution. This single-site study aims to enroll 50 participants.

ELIGIBILITY:
Inclusion Criteria:

* HIV-positive
* Between 30 and 70 years of age
* Elevated blood levels of fat
* On two or more anti-HIV drugs for at least12 months in a row and unlikely to change anti-HIV therapy during the study
* On stable regimen for at least 6 months for women taking oral contraceptive agents or hormone replacement
* On a stable regimen for at least 6 months for men on testosterone replacement
* If taking nevirapine, on therapy for at least 3 months with stable liver function tests

Exclusion Criteria:

* Pregnancy and breastfeeding
* Poorly controlled diabetes
* Uncontrolled hypertension or clinical evidence of heart failure
* Any serious medical conditions, including an active AIDS-defining condition, pancreatitis, or hepatitis within 6 months prior to the study
* Laboratory abnormalities (see investigator)
* On lipid lowering agents, insulin, anabolic steroids (except for testosterone at replacement doses), oral corticosteroids at greater than replacement doses, or growth hormones
* History of liver reaction or severe edema associated with current thiazolidinedione
* History of hypersensitivity to thiazolidinedione

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2003-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Carotid intima media thickness (IMT) | 1 year

SECONDARY OUTCOMES:
Changes in glucose metabolism | 1 year
Changes in concentrations of blood lipids | 1 year
Changes in C-reactive protein | 1 year
Changes in pre-inflammatory cytokines (MCP-1, IL-6) and adipocytokines (RBP-4, adiponectin) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Greg Bondy, MD, Principal Investigator — University of British Columbia
Locations (1):
- St. Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- See also: Related Info — http://www.hivnet.ubc.ca